CLINICAL TRIAL: NCT01258114
Title: Maâthermes a Randomised Controlled Trial of Spa Treatment of Overweight and Obesity
Brief Title: Maâthermes: Spa Treatment for Overweight and Obesity
Acronym: MAATHERMES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Association Francaise pour la Recherche Thermale (Other)
Collaborators: Université Joseph Fourier (Other); Université Victor Segalen Bordeaux 2 (Other); HAT Consultant (Unknown); AXONAL S.A. (Unknown)
Responsible Party: Docteur Renée-Claire MANCRET, Association Francaise pour la Recherche Thermale
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAATHERMES
Record Dates: First submitted 2010-12-08; First posted 2010-12-10 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity; Balneotherapy; Spa Therapy; balneology; hydrotherapy; SF 12; Nutritional counselling; Zelen double consent; Lifestyle modification program; IMC
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPA treatment (ST) (Active Comparator): Drug : spa treatment during 18 days soon after randomization the most adapted to the concerned pathology and common to all of spa resorts (mineral water drinking, bath with automatic air (bubble bathing), mud body wrapping, manual massages, water exercises) ;
  * nutritional counseling (french nutritional recommendations booklet) ;
  * caloric restriction and physical training on demand (non mandatory).
  Interventions: Other: SPA treatment (ST)
- Non SPA treatment (NST) (Sham Comparator): Drug: General practitioner (GP) counselling After randomisation Verbal and/or written advice based on the "French national guidelines for a healthy life style" brochure (given to the patient by the GP at baseline)
  Interventions: Other: Non SPA treatment (NST)

INTERVENTIONS:
Other: SPA treatment (ST) — Drug: spa treatment soon after randomization :
  Spa treatment of 18 days. Spa treatment : the most adapted to the concerned pathology and common to all of spa resorts (mineral water drinking, bath with automatic air (bubble bathing), mud body wrapping, manual massages, water exercises ;
  * nutritional counseling (french nutritional recommendations booklet) ;
  * caloric restriction and physical training on demand (non mandatory).
  Arms: SPA treatment (ST)
Other: Non SPA treatment (NST) — Drug: General practitioner (GP) counselling After randomisation Verbal and/or written advice based on the "French national guidelines for a healthy life style" brochure (given to the patient by the GP at baseline)
  Arms: Non SPA treatment (NST)

SUMMARY:
Public health campaigns and industry-supported changes in our food supply have obviously failed to control the epidemic to date. However, customized life style modification programs (LSMP) comprising diet, physical activity and behavioral therapy (a set of principles designed to help patients achieve their goals) induce weight loss of 10% of baseline body weight after 16 to 26 weeks of intervention . Long-term weight control is then facilitated by an appropriate weight-loss maintenance strategy such as continued patient-therapist contact (whether provided in person or by telephone or e-mail). This strategy allows patients to stabilize at an average of 5% and 3% loss of baseline body weight after 1 and 2 years, respectively. Numerous reports have concluded that this modest weight loss contributes to important health benefits.

However, the high dropout rate during weight-management strategies presumably means that treatment is mainly effective in highly motivated patients, as the highest success rates are likely to be reported among study completers. Many individuals appear to conclude that the benefits of weight-management strategies are not worth the cost (i.e. time, money, and continued unrewarding efforts). This underlines the critical need to implement new, practical and affordable strategies to induce and maintain weight loss that can be achieved by most patients.

The main objective of this study is to test the hypothesis that a 3 week intensive course of spa therapy can reduce the weight (and/or BMI) of overweight or obese patient at 14 months (BMI from 27 to 35).

DETAILED DESCRIPTION:
Spa therapy, or mineral spring water therapy, is a 3-week LSMP that has been shown to be sufficiently effective to control overweight and obesity to be approved and subsidized by French national health insurance. However, good quality scientific evidence is still required to support the benefit of spa therapy. An unpublished pilot study conducted in 2004, in several French spa resorts, showed that an additional 25% decrease in BMI was obtained for overweight and obese individuals enrolled in spa therapy as compared to individuals receiving classic weight management (-1.4 kg/m² and -1.05 kg/m2 respectively). However, no scientific conclusions can be drawn in the absence of relevant methodological and clinical information. This multicenter, controlled trial was designed to obtain sufficient statistical power to assess the benefits of spa therapy based on an evidence- based medicine approach.

The primary objective of this study was to assess whether a 3- week course of spa therapy is effective to achieve sustained weight loss over a period of 14 months among overweight and obese individuals

ELIGIBILITY:
Inclusion Criteria:

* Both sexes, more than 20 years and less than 70 years old patients with overweight (BMI>27) or obesity (BMI<35). Available for a spa treatment during 18 days, and a follow-up period of 14 months
* Voluntary to participate to the study,informed consent form signed after appropriate information
* Affiliation to the social security system or equivalent

Exclusion Criteria:

* Previous spa therapy for weight problems
* Pregnancy
* Major eating disorders (compulsive over eating)
* Poor french proficiency
* Involvement in another clinical trial
* Other contra-indications to spa therapy (severe general weakness, inflammatory bowel disease, cirrhosis, severe disability, psychosis and dementia, or Immunodeficiency, cancer in progress).
* Refusal to consent
* Refusal of spa treatment

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2007-03; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
SPA treatment (ST) : Active comparator spa treatment during 18 days soon after randomization. The Weight loss will be measured in kg and kg/m2 at 14 months | 14 months
  spa treatment during 18 days soon after randomization Weight loss assessed in kg and kg/m2 at 14 months

SECONDARY OUTCOMES:
Patients achieving a weight loss of 5% | 14 months
Quality of life : assessed by SF12 | 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick SEROG, MD, Principal Investigator — Hospital PARIS; Thierry HANH, MD, Study Director — PARIS HAT Consultant
Locations (5):
- France (5):
  - Cabinet Médical, Brides-les-Bains
  - Cabinet Medical, Capvern-les-Bains
  - Cabinet Medical, Vals-les-Bains
  - Cabinet Medical, Vichy
  - Cabinet Medical, Vittel

REFERENCES:
- [Background] Peneau S, Thibault H, Meless D, Soulie D, Carbonel P, Roinsol D, Longueville E, Serog P, Deheeger M, Bellisle F, Maurice-Tison S, Rolland-Cachera MF. Anthropometric and behavioral patterns associated with weight maintenance after an obesity treatment in adolescents. J Pediatr. 2008 May;152(5):678-84. doi: 10.1016/j.jpeds.2007.09.053. Epub 2007 Nov 26. PMID 18410773
- [Background] Rolland-Cachera MF, Thibault H, Souberbielle JC, Soulie D, Carbonel P, Deheeger M, Roinsol D, Longueville E, Bellisle F, Serog P. Massive obesity in adolescents: dietary interventions and behaviours associated with weight regain at 2 y follow-up. Int J Obes Relat Metab Disord. 2004 Apr;28(4):514-9. doi: 10.1038/sj.ijo.0802605. PMID 14968129
- [Background] Marcellin P, Cadranel JF, Fontanges T, Poynard T, Pol S, Trepo C, Blin P, Bregman B, Schmidely N, Roudot-Thoraval F, Zarski JP. High rate of adefovir-lamivudine combination therapy in nucleoside-naive patients with chronic hepatitis B in France: results of a national survey in 1730 patients. Eur J Gastroenterol Hepatol. 2010 Nov;22(11):1290-6. doi: 10.1097/meg.0b013e32832fba4f. PMID 20964259
- [Background] Fourrier-Reglat A, Lacoin L, Pariente A, Lassalle R, Robinson P, Droz-Perroteau C, Begaud B, Blin P, Moore ND. When patients report diseases that prescribers seem unaware of: discordance between patient and physician reporting of risk-related previous history in NSAID users from the CADEUS study. Clin Pharmacol Ther. 2010 Nov;88(5):668-75. doi: 10.1038/clpt.2010.166. Epub 2010 Sep 22. PMID 20861835
- [Background] Blin P, Blazejewski S, Lignot S, Lassalle R, Bernard MA, Jayles D, Theophile H, Benichou J, Demeaux JL, Ebbo D, Franck J, Moride Y, Peyramond D, Rouveix B, Sturkenboom M, Gehanno P, Droz C, Moore N. Effectiveness of antibiotics for acute sinusitis in real-life medical practice. Br J Clin Pharmacol. 2010 Sep;70(3):418-28. doi: 10.1111/j.1365-2125.2010.03710.x. PMID 20716243
- [Background] Saraux A, Combe B, Blin P, Bregman B, Chartier M, Durieux-Mehlman S, Guillemin F. Survey of the therapeutic management of rheumatoid arthritis in France: the OPALE study. Clin Exp Rheumatol. 2010 May-Jun;28(3):325-32. Epub 2010 Jun 23. PMID 20460034
- [Background] Fourrier-Reglat A, Cuong HM, Lassalle R, Depont F, Robinson P, Droz-Perroteau C, Pariente A, Begaud B, Blin P, Moore N. Concordance between prescriber- and patient-reported previous medical history and NSAID indication in the CADEUS cohort. Pharmacoepidemiol Drug Saf. 2010 May;19(5):474-81. doi: 10.1002/pds.1951. PMID 20437457
- [Background] Colver AF, Dickinson HO; SPARCLE group. Study protocol: determinants of participation and quality of life of adolescents with cerebral palsy: a longitudinal study (SPARCLE2). BMC Public Health. 2010 May 26;10:280. doi: 10.1186/1471-2458-10-280. PMID 20504349
- [Background] Colver AF, Dickinson HO, Parkinson K, Arnaud C, Beckung E, Fauconnier J, Marcelli M, McManus V, Michelsen SI, Parkes J, Thyen U. Access of children with cerebral palsy to the physical, social and attitudinal environment they need: a cross-sectional European study. Disabil Rehabil. 2011;33(1):28-35. doi: 10.3109/09638288.2010.485669. Epub 2010 May 6. PMID 20446803
- [Background] Fauconnier J, Pasquie JL, Bideaux P, Lacampagne A, Richard S. Cardiomyocytes hypertrophic status after myocardial infarction determines distinct types of arrhythmia: role of the ryanodine receptor. Prog Biophys Mol Biol. 2010 Sep;103(1):71-80. doi: 10.1016/j.pbiomolbio.2010.01.002. Epub 2010 Jan 28. PMID 20109482
- [Background] Fauconnier J, Thireau J, Reiken S, Cassan C, Richard S, Matecki S, Marks AR, Lacampagne A. Leaky RyR2 trigger ventricular arrhythmias in Duchenne muscular dystrophy. Proc Natl Acad Sci U S A. 2010 Jan 26;107(4):1559-64. doi: 10.1073/pnas.0908540107. Epub 2010 Jan 4. PMID 20080623
- [Background] Casez P, Labarere J, Sevestre MA, Haddouche M, Courtois X, Mercier S, Lewandowski E, Fauconnier J, Francois P, Bosson JL. ICD-10 hospital discharge diagnosis codes were sensitive for identifying pulmonary embolism but not deep vein thrombosis. J Clin Epidemiol. 2010 Jul;63(7):790-7. doi: 10.1016/j.jclinepi.2009.09.002. Epub 2009 Dec 2. PMID 19959332
- [Background] Mansen A, Tiselius C, Sand P, Fauconnier J, Westerblad H, Rydqvist B, Vennstrom B. Thyroid hormone receptor alpha can control action potential duration in mouse ventricular myocytes through the KCNE1 ion channel subunit. Acta Physiol (Oxf). 2010 Feb;198(2):133-42. doi: 10.1111/j.1748-1716.2009.02052.x. Epub 2009 Oct 14. PMID 19832729
- [Background] Messing B, Man F, Therond P, Hanh T, Thuillier F, Rambaud JC. Selenium status prior to and during one month total parenteral nutrition in gastroenterological patients: A randomised study of two dosages of Se supplementation. Clin Nutr. 1990 Oct;9(5):281-8. doi: 10.1016/0261-5614(90)90037-s. PMID 16837371